CLINICAL TRIAL: NCT06663241
Title: Validation of New Photographic Technology for Assessing Skin Lesions
Brief Title: The Validation of New Photographic Technology for Assessing Skin Lesions
Status: Completed | Type: Observational
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-2022-151
Record Dates: First submitted 2024-10-18; First posted 2024-10-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Skin Lesions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

SUMMARY:
The purpose of this study is to determine the validity of a new photographic technology in a dermatologic setting. The digital picture uses high levels of resolution to look at skin biopsy lesions. These photos will be compared to current standard-of-care with hematoxylin and eosin histologic analysis by board-certified dermatologists.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ages 18 and older.
* Able to comprehend procedures, risks, and informed consent.
* Have a skin lesion the practitioner believes, and subject agrees, should be biopsied.
* Lesion on a non-revealing part of the body (none on areas that would be recognizable, nor on groin nor breasts).
* Willingness of subject to share the results of the biopsy pathology.

Exclusion Criteria:

* Lesion on a revealing part of body.
* Unable to understand the procedures, informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wright State Physicians Dermatology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Number of matching dermatologic diagnoses from photography to biopsied lesions. | At time of biopsy procedure of the lesion.
  A group of board-certified dermatologists will evaluate the standard digital vs. enhanced digital photograph of the lesion to compare the accuracy of diagnoses to the pathology report, with pathology serving as the gold standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States

IPD SHARING:
Plan to Share IPD: No